CLINICAL TRIAL: NCT03169907
Title: Cardiac Functions as a New Method for Evaluation of Fetal Anemia Pre and Post Intrauterine Fetal Blood Transfusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre, Egypt (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NRC-002
Record Dates: First submitted 2017-02-21; First posted 2017-05-30 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2017-05

CONDITIONS: Fetal Anemia as Antepartum Condition (Diagnosis); Rh Incompatible Blood Transfusion Nos
Keywords: Cardiac functions; Intrauterine fetal anemia; Intrauterine Fetal blood transfusion; Myocardial performance index; spatiotemporal imaging correlation
MeSH Terms: conditions — Disease

STUDY DESIGN:
Intervention Model Description: This will be a prospective study. Patients will be selected from Rh isoimmunized patients (positive titre of indirect coomb's test) who are scheduled to have intrauterine blood transfusion.Selected patients will be monitored weekly from 15 weeks gestational age till 28 weeks of gestational age.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rh isoimmunized patients (Experimental): Patients will be selected from Rh isoimmunized patients (positive titre of indirect coomb's test) who are scheduled to have intrauterine blood transfusion. This intrauterine blood transfusion is due to fetal anemia, and it is detected when the measurement of PSV (peak systolic velocity) of middle cerebral artery is more than 1.5 MoM (multiple of the median) according to Fetal Medicine unit of Cairo University protocol. All fetuses are free of structural and functional Fetal and echocardiographic anomaly scan.
  Interventions: Radiation: Mid trimesteric fetal ultrasonography

INTERVENTIONS:
Radiation: Mid trimesteric fetal ultrasonography — Venous and arterial Doppler indices:
  1. Middle cerebral artery (MCA) peak systolic velocity (PSV):
  2. Umbilical Artery Pulsitility Index (PI) and Resistant Index (RI):
  3. Ductus venosus (DV) Doppler:
  Cardiac functions:
  1. Global cardiac function evaluated by Modified Myocardial Performance Index (Mod-MPI):
  2. Systolic cardiac function using the four-dimensional (4D) spatiotemporal imaging correlation (STIC) ultrasound technique:
  3. Diastolic cardiac function evaluated by relationship between the maximal velocities of the E and A waveforms of ventricular filling (E/A ratio)
  Other Names: Voluson E10 equipment (GE Medical Systems, Austria)

SUMMARY:
INTRODUCTION

Circulatory changes associated with fetal anemia have an important role in maintaining sufficient tissue oxygenation. With fetal anemia, hyperdynamic circulation and increased cardiac output occurred. In current practice, using Doppler in assessment of the peak systolic velocity (PSV) of the middle cerebral artery (MCA) is the main parameter in screening of fetal anemia. Myocardial performance index (MPI) is a noninvasive technique that evaluates systolic and diastolic cardiac function by pulsed Doppler.

Patients and Methods:

This prospective study will be carried out on Women with singleton pregnancies with Rh isoimmunization who are scheduled to have intrauterine blood transfusion. Selected patients will be monitored weekly from 18 weeks gestational age till 28 weeks of gestational age.

Venous and arterial Doppler indices:

1. Middle cerebral artery (MCA) peak systolic velocity (PSV)
2. Umbilical Artery Pulsitility Index (PI) and Resistant Index (RI)
3. Ductus venosus (DV) Doppler

Cardiac functions:

1. Global cardiac function evaluated by Modified Myocardial Performance Index (Mod-MPI)
2. Diastolic cardiac function evaluated by relationship between the maximal velocities of the E and A waveforms of ventricular filling (E/A ratio)

DETAILED DESCRIPTION:
INTRODUCTION

Circulatory changes associated with fetal anemia have an important role in maintaining sufficient tissue oxygenation. With fetal anemia, hyperdynamic circulation and increased cardiac output occurred. This is due to reduced the viscosity of blood, increased the contractility of heart, and peripheal vasodilatation due to hypoxia. In current practice, using Doppler in assessment of the peak systolic velocity (PSV) of the middle cerebral artery (MCA) is the main parameter in screening of fetal anemia. Severe fetal anemia causes continuous loss of adaptive mechanisms due to lack of oxygen delivered to the tissues. Finally, fetal acidosis results as a sequence of metabolic changes so increasing perinatal morbidity and mortality. Cardiac decompensation is not the principal mechanism involved in the development of overt fetal hydrops, however, severe anemia may cause cardiac ischemia, reduced contractility, and dysfunction. Myocardial performance index (MPI) is a noninvasive technique that evaluates systolic and diastolic cardiac function by pulsed Doppler. Tsutsumi et al. was the first described Fetal MPI evaluation then several studies have shown that it is a simple and replicable technique. Many have demonstrated significant changes in fetal MPI in intrauterine growth restriction, recipient fetuses of twin-twin transfusion syndrome, diabetes, and fetal inflammatory response syndrome. Similarly, fetal anemia causes changes in cardiac contractility and MPI as one of cardiac functions may have a role in the evaluation of disease severity and prognosis.

Patients and Methods:

This prospective study will be carried out at a tertiary referral center for fetal medicine (Fetal Medicine Unit, Cairo University, Egypt) from April 2017 till April 2018. Women with singleton pregnancies with Rh isoimmunization will be asked to participate in the study. Informed consent will be obtained from all participants. The ethical committee approval for the study will be from Bioethical Committee of the National Research Centre (number: 17 008, admission date: January 2017).

This will be a prospective study. Patients will be selected from Rh isoimmunized patients (positive titer of indirect coomb's test) who are scheduled to have intrauterine blood transfusion. This intrauterine blood transfusion is due to fetal anemia, and it is detected when the measurement of PSV (peak systolic velocity) of middle cerebral artery is more than 1.5 MoM (multiple of the median) according to Fetal Medicine unit of Cairo University protocol. All fetuses are free of structural and functional Fetal and echocardiographic anomaly scan.

Gestational age will be obtained from the first date of the last menstrual period (LMP). If the patient is unsure of her dates, gestational age will be based on the first ultrasound scan. Selected patients will be monitored weekly from 18 weeks gestational age till 28 weeks of gestational age.

All examinations will be carried out abdominally with a curved 3.5-5.0-MHz probe and Voluson E10 equipment (General Electric Medical Systems, Austria). Data will be entered into an electronic spreadsheet (Excel,Microsoft Corporation, USA).

Fetal Hemoglobin (Hb) levels will be measured in blood samples collected prior to transfusion and after blood transfusion before withdrawing of the needle from umbilical vein.

Venous and arterial Doppler indices:

1. Middle cerebral artery (MCA) peak systolic velocity (PSV):

   The greatest measurement of three consequent PSV will be recorded. the course of the fetal MCA will be identified by using color Doppler. An axial brain section of the fetus, including the thalami and the cavitas septi pellucid (CSP), will be obtained. And the MCA will be captured along the great wing of the sphenoid bone. The artery will be examined close to its origin with angle of insonation < 20 degrees.
2. Umbilical Artery Pulsitility Index (PI) and Resistant Index (RI):

   Both umbilical arteries will be sampled close to the placental insertion and ultrasound 3.5-5-MHz convex probes will be used, the insonation angle will be <30° and the sample volume will be adjusted to cover the entire vessel.
3. Ductus venosus (DV) Doppler:

The flow velocities from the DV will be identified using color Doppler imaging in a right ventral midsagittal plane. The pulsed Doppler gate will be placed in the distal portion of the umbilical sinus. When the typical DV waveform is obtained, at least three consecutive waveforms will be recorded with insonation angle < 30. The following variables will be measured: S-wave, D-wave, pulsatility index for veins (PIV) and resistance index (RI).

Cardiac functions:

1. Global cardiac function evaluated by Modified Myocardial Performance Index (Mod-MPI):

   All estimations will be done in the absence of fetal corporal and respiratory movements and with the mother in voluntary suspended respiration. Special attention will be given to the velocity of the Doppler sweep representation on the ultrasound screen using the highest velocity available (15 cm/s) for clear identification of the components of the Doppler tracing. Additionally, the E/A waveform will always be displayed as positive flow. The angle of insonation will always be kept below 30◦ and the mechanical and thermal indices will never exceeded 1. A cross-sectional image of the fetal thorax in the four-chamber view and an apical projection of the heart will be obtained. The Doppler sample volume will be placed on the lateral wall of the ascending aorta, below the AV (aortic valve) and just above the MV (mitral valve). The Doppler trace will show a clear echo corresponding to the opening and closure of the two valves at the beginning and at the end of the E/A (mitral valve) and AF (aortic flow) waveforms. The time periods will then be estimated as follows: the isovolumetric contraction time (ICT) will be estimated from the closure of the MV, to the opening of the AV, the ET (ejection time) from the opening to the closure of the AV, and the IRT (the isovolumetric relaxation time ) from the closure of the AV to the opening of the MV. The final value for the Mod-MPI will be calculated as: (ICT+IRT)/ET.
2. Systolic cardiac function using the four-dimensional (4D) spatiotemporal imaging correlation (STIC) ultrasound technique:

   Fetal heart ventricular volumes will be measured using the four-dimensional (4D) spatiotemporal imaging correlation (STIC) ultrasound technique. TheVirtual Organ Computer-aided AnaLysis (VOCAL) technique will be used to obtain a sequence of six sections of each ventricular volume in systole and diastole. Each volume will be obtained after a 60 degree rotation from the previous one around a fixed axis extending from the apex of the heart to the point that divides symmetrically each atrioventricular valve. The contour of each ventricle will be drawn manually and the 4D volumes of the left and right ventricle in systole and diastole will be estimated. The stroke volume for each ventricle will then be calculated by subtracting the one in systole from the one in diastole and the cardiac output will be calculated by multiplying the stroke volume by the fetal heart rate.
3. Diastolic cardiac function evaluated by relationship between the maximal velocities of the E and A waveforms of ventricular filling (E/A ratio):

Assessment of the fetal diastolic component of the cardiac cycle is performed with spectral Doppler through the atrioventricular (AV) valves. The Doppler sample gate is located just below the AV valves where a biphasic waveform is usually displayed in normal fetus and is kept gate between 2 and 3 mm. The first component is known as the E (early or passive) wave and is related to the process of myocardial relaxation and negative pressure applied by the ventricles. The second component is the A (atrial, active, or late) wave and it represents the atrial contraction during ventricular filling. The ratio is obtained by the division of the peak velocities of the E over the A waveforms. Recordings are obtained at the level of the 4-chamber view of the fetal heart in either a posterior or an anterior apical projection. The interventricular septum must be visualized and aligned at 0 degree with the Doppler beam and angle of insonation < 20 degrees.

ELIGIBILITY:
Inclusion Criteria:

* Rh isoimmunized patients (positive titre of indirect coomb's test) who are scheduled to have intrauterine blood transfusion.

Exclusion Criteria:

* Less than 15 weeks gestational age and more than 28 weeks gestational age
* fetuses with structural or functional Fetal or echocardiographic anomalies.

Ages: 18 Weeks to 28 Weeks | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Modified Myocardial Performance Index (Mod-MPI) | 10 seconds
  the ratio between summation of isovolumetric contraction time (ICT) + isovolumetric relaxation time (IRT) in melliseconds and ejection time (ET) in melliseconds

SECONDARY OUTCOMES:
Fetal Hemoglobin (Hb) levels | 15 minutes
  Fetal Hemoglobin (Hb) levels which is measured by g/dl. A blood sample is collected from umbilical vein prior to blood transfusion (Sample 1) and another blood sample (Sample 2) after blood transfusion just before withdrawing of the trnsfusion needle from umbilical vein
Middle cerebral artery (MCA) peak systolic velocity (PSV) | 10 seconds
  MCA PSV will be identified by using pulsed wave Doppler in cm/s
(E/A) ratio | 10 seconds
  The relationship between the maximal velocities of the E and A waveforms of ventricular filling

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Z El Sheikhah, Professor, Principal Investigator — Professor of Obstetrics and Gynecology, Cairo Fetal Medicine Unit, Cairo University
Locations (1):
- Cairo University, Faculty of Medicine, Obstetrics and Gynecology Department, Cairo Fetal Medicine Unit., Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bilardo CM, Nicolaides KH, Campbell S. Doppler studies in red cell isoimmunization. Clin Obstet Gynecol. 1989 Dec;32(4):719-27. doi: 10.1097/00003081-198912000-00013. No abstract available. PMID 2515021
- [Background] Nicolaides KH. Studies on fetal physiology and pathophysiology in rhesus disease. Semin Perinatol. 1989 Aug;13(4):328-37. No abstract available. PMID 2528210
- [Background] Hecher K, Snijders R, Campbell S, Nicolaides K. Fetal venous, arterial, and intracardiac blood flows in red blood cell isoimmunization. Obstet Gynecol. 1995 Jan;85(1):122-8. doi: 10.1016/0029-7844(94)00331-7. PMID 7800308
- [Background] Mari G, Deter RL, Carpenter RL, Rahman F, Zimmerman R, Moise KJ Jr, Dorman KF, Ludomirsky A, Gonzalez R, Gomez R, Oz U, Detti L, Copel JA, Bahado-Singh R, Berry S, Martinez-Poyer J, Blackwell SC. Noninvasive diagnosis by Doppler ultrasonography of fetal anemia due to maternal red-cell alloimmunization. Collaborative Group for Doppler Assessment of the Blood Velocity in Anemic Fetuses. N Engl J Med. 2000 Jan 6;342(1):9-14. doi: 10.1056/NEJM200001063420102. PMID 10620643
- [Background] Moise KJ Jr, Mari G, Fisher DJ, Huhta JC, Cano LE, Carpenter RJ Jr. Acute fetal hemodynamic alterations after intrauterine transfusion for treatment of severe red blood cell alloimmunization. Am J Obstet Gynecol. 1990 Sep;163(3):776-84. doi: 10.1016/0002-9378(90)91067-m. PMID 2119560
- [Background] Tongsong T, Tongprasert F, Srisupundit K, Luewan S. Venous Doppler studies in low-output and high-output hydrops fetalis. Am J Obstet Gynecol. 2010 Nov;203(5):488.e1-6. doi: 10.1016/j.ajog.2010.06.003. Epub 2010 Aug 3. PMID 20684946
- [Background] Tei C, Ling LH, Hodge DO, Bailey KR, Oh JK, Rodeheffer RJ, Tajik AJ, Seward JB. New index of combined systolic and diastolic myocardial performance: a simple and reproducible measure of cardiac function--a study in normals and dilated cardiomyopathy. J Cardiol. 1995 Dec;26(6):357-66. PMID 8558414
- [Background] Tsutsumi T, Ishii M, Eto G, Hota M, Kato H. Serial evaluation for myocardial performance in fetuses and neonates using a new Doppler index. Pediatr Int. 1999 Dec;41(6):722-7. doi: 10.1046/j.1442-200x.1999.01155.x. PMID 10618901
- [Background] Eidem BW, Edwards JM, Cetta F. Quantitative assessment of fetal ventricular function: establishing normal values of the myocardial performance index in the fetus. Echocardiography. 2001 Jan;18(1):9-13. doi: 10.1046/j.1540-8175.2001.t01-1-00009.x. PMID 11182775
- [Background] Friedman D, Buyon J, Kim M, Glickstein JS. Fetal cardiac function assessed by Doppler myocardial performance index (Tei Index). Ultrasound Obstet Gynecol. 2003 Jan;21(1):33-6. doi: 10.1002/uog.11. PMID 12528158
- [Background] Ichizuka K, Matsuoka R, Hasegawa J, Shirato N, Jimbo M, Otsuki K, Sekizawa A, Farina A, Okai T. The Tei index for evaluation of fetal myocardial performance in sick fetuses. Early Hum Dev. 2005 Mar;81(3):273-9. doi: 10.1016/j.earlhumdev.2004.07.003. PMID 15814209
- [Background] Szwast A, Tian Z, McCann M, Donaghue D, Bebbington M, Johnson M, Wilson RD, Rychik J. Impact of altered loading conditions on ventricular performance in fetuses with congenital cystic adenomatoid malformation and twin-twin transfusion syndrome. Ultrasound Obstet Gynecol. 2007 Jul;30(1):40-6. doi: 10.1002/uog.4032. PMID 17533619
- [Background] Crispi F, Hernandez-Andrade E, Pelsers MM, Plasencia W, Benavides-Serralde JA, Eixarch E, Le Noble F, Ahmed A, Glatz JF, Nicolaides KH, Gratacos E. Cardiac dysfunction and cell damage across clinical stages of severity in growth-restricted fetuses. Am J Obstet Gynecol. 2008 Sep;199(3):254.e1-8. doi: 10.1016/j.ajog.2008.06.056. PMID 18771973
- [Background] Letti Muller AL, Barrios Pde M, Kliemann LM, Valerio EG, Gasnier R, Magalhaes JA. Tei index to assess fetal cardiac performance in fetuses at risk for fetal inflammatory response syndrome. Ultrasound Obstet Gynecol. 2010 Jul;36(1):26-31. doi: 10.1002/uog.7584. PMID 20131338
- [Background] Van Mieghem T, Gucciardo L, Lewi P, Lewi L, Van Schoubroeck D, Devlieger R, De Catte L, Verhaeghe J, Deprest J. Validation of the fetal myocardial performance index in the second and third trimesters of gestation. Ultrasound Obstet Gynecol. 2009 Jan;33(1):58-63. doi: 10.1002/uog.6238. PMID 18973212
- [Background] de Assuncao RA, Liao AW, de Lourdes Brizot M, Francisco RP, Zugaib M. Myocardial performance index in fetal anemia. Prenat Diagn. 2015 Feb;35(2):192-6. doi: 10.1002/pd.4526. Epub 2014 Dec 15. PMID 25377887
- [Background] Nishie EN, Brizot ML, Liao AW, Carvalho MH, Toma O, Zugaib M. A comparison between middle cerebral artery peak systolic velocity and amniotic fluid optical density at 450 nm in the prediction of fetal anemia. Am J Obstet Gynecol. 2003 Jan;188(1):214-9. doi: 10.1067/mob.2003.63. PMID 12548220
- [Background] Tseng CC, Wang HI, Wang PH, Yang MJ, Juang CM, Horng HC, Wu YC, Chen CC, Shiu HL, Chiang MM, Lin HJ, Chen CY, Chao KC. Ductus venosus Doppler velocimetry in normal pregnancies from 11 to 13 + 6 weeks' gestation - a Taiwanese study. J Chin Med Assoc. 2012 Apr;75(4):171-5. doi: 10.1016/j.jcma.2012.02.015. Epub 2012 Mar 31. PMID 22541146
- [Background] Hernandez-Andrade E, Lopez-Tenorio J, Figueroa-Diesel H, Sanin-Blair J, Carreras E, Cabero L, Gratacos E. A modified myocardial performance (Tei) index based on the use of valve clicks improves reproducibility of fetal left cardiac function assessment. Ultrasound Obstet Gynecol. 2005 Sep;26(3):227-32. doi: 10.1002/uog.1959. PMID 16116562